CLINICAL TRIAL: NCT04080791
Title: Efficacy of Virtual Reality in Stroke Rehabilitation
Brief Title: Virtual Reality in Stroke Rehabilitation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00052687
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Ischemic Stroke
Keywords: Virtual Reality; Stroke; National Stroke Association; Stroke Rehabilitation
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Drug Delivery Systems; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental Group- Virtual Reality (VR) Treatment (Experimental): The participants in the experimental group will complete the educational/training session on how to use the VR equipment and programs (30 minutes). The following day, participants will begin the VR intervention attending a daily 30-minute sessions for 8 days or until a discharge date has been set, whichever comes first.
  Interventions: Device: Virtual Reality (VR) System; Procedure: Standard of care
- Standard of care group (Active Comparator): The control group participants will receive the traditional daily 30-minute intensive therapy regimen provided during acute inpatient rehabilitation stroke treatment protocol. Prior to discharge, control group participants will meet with a licensed clinical therapist to complete the cognitive and physical assessments for the posttest evaluation.
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Device: Virtual Reality (VR) System — The participants will undergo daily 30-minute sessions for 8 days of Virtual Reality (VR) with a VR system using commercially available default programs in addition to traditional intensive therapy regimen provided during inpatient rehab.
  Arms: Experimental Group- Virtual Reality (VR) Treatment
Procedure: Standard of care — Control group participants will receive the traditional daily 30-minute intensive therapy regimen provided during acute inpatient rehabilitation stroke treatment protocol.

SUMMARY:
The purpose of this research study is to investigate the effects of Virtual Reality (VR) as a treatment intervention to increase physical and cognitive function in stroke survivors.

DETAILED DESCRIPTION:
In this pilot study, the objective is to determine if there is an increase in MoCA (Montreal Cognitive Assessment), MFRT (Modified Functional Reach Test), and FMA-UA (Fugl-Meyer Assessment Upper Extremity) scores of participants who receive the VR intervention in addition to traditional inpatient rehabilitation standard of care (experimental group) versus participants who receive the traditional standard of care (control group).

ELIGIBILITY:
Inclusion Criteria:

* Patients Age 18 and older admitted to inpatient rehabilitation with a projected LOS (length of stay) of 10 days or more within the open data collection period for treatment of ischemic stroke and agree to participate in the study in addition to traditional intensive rehabilitation therapy.

Exclusion Criteria:

* Individual patients who exhibit the following symptoms or medical history or are not medically cleared for participation will be excluded:
* History of, or high risk for, seizures
* Feed tube, tracheotomy, or other medical devices that would preclude the use or wear of the VR headset as it covers the face and head
* Blindness
* History of mental health issues such as schizophrenia, manic episodes, active psychosis, or other mental health issues that may be exacerbated by exposure to VR
* Open wounds that would preclude use for the VR headset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | baseline
  Scores range from 0 to 30 with higher scores denoting better outcomes.
Montreal Cognitive Assessment (MoCA) | Up to 8 days after baseline
  Scores range from 0 to 30 with higher scores denoting better outcomes.
Modified Functional Reach Test (MFRT) | baseline
  The Modified Functional Reach Test will be used to measure physical functioning. Measurements are the maximum distance the patient can reach forward while sitting in a fixed position. A score of 6 or less indicates a significant increased risk of falls. A score between 6-10 inches indicates a moderate risk for falls.
Modified Functional Reach Test (MFRT) | Up to 8 days after baseline
  The Modified Functional Reach Test will be used to measure physical functioning. Measurements are the maximum distance the patient can reach forward while sitting in a fixed position. A score of 6 or less indicates a significant increased risk of falls. A score between 6-10 inches indicates a moderate risk for falls.
FMA-UE (Fugl-Meyer Assessment for Upper Extremity) | baseline
  Fugl-Meyer Assessment for Upper Extremity will be used to measure upper extremity motor function. Scores range from 0 (unable to do the task) to 66 (task performed fully). Higher scores denote better outcome.
FMA-UE (Fugl-Meyer Assessment for Upper Extremity) | Up to 8 days after baseline
  Fugl-Meyer Assessment for Upper Extremity will be used to measure upper extremity motor function. Scores range from 0 (unable to do the task) to 66 (task performed fully). Higher scores denote better outcome.

SECONDARY OUTCOMES:
Pain intensity self-report ratings | prior to VR treatment, day 1, and days 2, 3, 4, 5, 6, 7, and 8 after baseline
  For subjects randomized into VR group only. Scores range from 0 to 10. Higher scores denote more pain intensity.
Pain intensity self-report ratings | immediately after VR treatment, day 1 and days 2, 3, 4, 5, 6, 7, and 8 after baseline
  For subjects randomized into VR group only. Scores range from 0 to 10. Higher scores denote more pain intensity.
Wong-Baker FACES scale | prior to VR treatment, day 1 and days 2, 3, 4, 5, 6, 7, and 8 after baseline
  For subjects randomized into VR group only. Scores range from 0 to 10. Higher scores denote more pain intensity.
Wong-Baker FACES scale | immediately after VR treatment, day 1 and days 2, 3, 4, 5, 6, 7, and 8 after baseline
  For subjects randomized into VR group only. Scores range from 0 to 10. Higher scores denote more pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Cromer, LRT, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henderson A, Korner-Bitensky N, Levin M. Virtual reality in stroke rehabilitation: a systematic review of its effectiveness for upper limb motor recovery. Top Stroke Rehabil. 2007 Mar-Apr;14(2):52-61. doi: 10.1310/tsr1402-52. PMID 17517575
- [Background] National Stroke Association, (2018) Stroke 101: Fast facts on stroke, accessed from url http://www.stroke.org/sites/default/files/resources/NSA_%20FactSheet_Strok e_101_2014.pdf
- [Background] Turolla A, Dam M, Ventura L, Tonin P, Agostini M, Zucconi C, Kiper P, Cagnin A, Piron L. Virtual reality for the rehabilitation of the upper limb motor function after stroke: a prospective controlled trial. J Neuroeng Rehabil. 2013 Aug 1;10:85. doi: 10.1186/1743-0003-10-85. PMID 23914733
- [Background] IBM Corp. (2012). IBM SPSS Statistics for Windows, Version 21.0. Armonk, NY: IBM Corp